CLINICAL TRIAL: NCT03770936
Title: Clinical Study Evaluating the Efficacy of Renin Angiotensin System Inhibitors on the Extent of Liver Fibrosis in Patients With Chronic Hepatitis C
Brief Title: Effect of Some Drugs on Liver Fibrosis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sherief Abd-Elsalam (Other)
Responsible Party: Sponsor-Investigator, Sherief Abd-Elsalam, Ass. Prof. Tropical Medicine, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: liver fibrosis
Record Dates: First submitted 2018-12-07; First posted 2018-12-10 (Actual); Last update posted 2018-12-10 (Actual); Status verified 2018-12

CONDITIONS: Liver Fibroses
MeSH Terms: conditions — Liver Cirrhosis | interventions — candesartan; Ramipril

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): No intervention
- Candesartan (Active Comparator): Candesartan 8 mg/day
  Interventions: Drug: Candesartan
- Ramipril (Active Comparator): Ramipril 1.25 mg/day
  Interventions: Drug: Ramipril

INTERVENTIONS:
Drug: Candesartan — Candesartan 8 mg/day
  Other Names: Cansartan
  Arms: Candesartan
Drug: Ramipril — ramipril 1.25 mg/day
  Arms: Ramipril

SUMMARY:
Effect of Some Drugs on Liver Fibrosis

DETAILED DESCRIPTION:
The study aimed at evaluating the effect of Some Drugs on Liver Fibrosis

ELIGIBILITY:
Inclusion Criteria:

* chronic hepatitis C

Exclusion Criteria:

* Acute hepatitis
* Thalassemia

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Change in Fibroscan or APRI score | 6 months
  Change in Fibroscan or APRI score

CONTACTS AND LOCATIONS:
Overall Officials: Gamal El-azab, Prof, Principal Investigator — Clinical pharmacy Department- Tanta University; Tarek Mostafa, Prof, Study Director — Cardiology Department- Tanta University; Gamal Badra, Prof, Study Chair — National Hepatology Institute - Egypt; Abeer El-Motwally, Msc, Study Chair — Clinical pharmacy Department-Tanta University
Locations (1):
- Sherief Abd-Elsalam, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mostafa TM, El-Azab GA, Badra GA, Abdelwahed AS, Elsayed AA. Effect of Candesartan and Ramipril on Liver Fibrosis in Patients with Chronic Hepatitis C Viral Infection: A Randomized Controlled Prospective Study. Curr Ther Res Clin Exp. 2021 Nov 12;95:100654. doi: 10.1016/j.curtheres.2021.100654. eCollection 2021. PMID 34925649